CLINICAL TRIAL: NCT02772653
Title: Evaluation of Resuscitation Markers in Trauma Patients
Status: Completed | Type: Observational
Sponsor: Andrea Campos-Serra (Other)
Collaborators: Corporacion Parc Tauli (Other)
Responsible Party: Sponsor-Investigator, Andrea Campos-Serra, MD, Corporacion Parc Tauli
Organization: Corporacion Parc Tauli (Other)
Other Study IDs: CSPT-CG-PPT1
Record Dates: First submitted 2016-05-07; First posted 2016-05-13 (Estimated); Last update posted 2019-05-14 (Actual); Status verified 2019-05

CONDITIONS: Trauma; Hypovolemic Shock
Keywords: Microcirculation; Videomicroscopy; Spectroscopy, Near-Infrared; B-Type Natriuretic Peptide; Thromboelastometry; Trauma; Resuscitation; Hypovolemic shock
MeSH Terms: conditions — Wounds and Injuries; Shock | interventions — Spectroscopy, Near-Infrared

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood samples for Natriuretic Peptide analysis. Retained just for one month, until samples are analyzed at an external laboratory.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Severe trauma patients: No interventions are done. It's a prospective and descriptive observational study where different markers are analyzed:
  * Blood Lactate levels
  * Blood Base Excess levels
  * Blood B-type Natriuretic Peptide levels
  * Blood Thromboelastometry (ROTEM) alterations
  * Near-infrared spectroscopy alterations
  * Sublingual videomicroscopy alterations
  All these markers are analyzed at the 1rst, 8th and 24th hour from hospital admission.
  Interventions: Other: Blood Lactate; Other: Blood Base Excess; Other: Blood B-type Natriuretic Peptide; Other: Blood Thromboelastometry (ROTEM); Other: Near-infrared spectroscopy; Other: Sublingual videomicroscopy

INTERVENTIONS:
Other: Blood Lactate — Analyzed at the 1rst, 8th and 24th hour from hospital admission
Other: Blood Base Excess — Analyzed at the 1rst, 8th and 24th hour from hospital admission
Other: Blood B-type Natriuretic Peptide — Analyzed at the 1rst, 8th and 24th hour from hospital admission
Other: Blood Thromboelastometry (ROTEM) — Analyzed at the 1rst, 8th and 24th hour from hospital admission
Other: Near-infrared spectroscopy — Analyzed at the 1rst, 8th and 24th hour from hospital admission
Other: Sublingual videomicroscopy — Analyzed at the 1rst, 8th and 24th hour from hospital admission

SUMMARY:
Severe trauma patients have an elevated risk of multiple organ failure and death. In order to increase survival possibilities the initial treatment must be focused into resuscitation from shock. Traditionally the most common resuscitation markers used are vital signs and urine output. Unfortunately, many patients might present normal vital signs, but still undergo a compensated shock with persistent acidosis, hence being able to develop multiple organ failure and death. Consequently, it is important to define better resuscitation markers for these patients.

This investigation project consists in an observational prospective study, performed by a multidisciplinary team, in which different resuscitation markers are evaluated in severe trauma patients. There will be a specific timing (1st, 8th and 24th hours from arrival) evaluation of different markers: hemodynamic (vital signs, urine output, etc); analytical (lactate, base excess, natriuretic atrial peptide); tissue perfusion markers (NIRS); microcirculation markers (videomicroscopy) and coagulopathy markers (thromboelastometry). There will be a registry of total volume administration; blood cell transfusions and vasoactive drug requirements. Each marker will be evaluated in relation to mortality; multiple organ failure; massive transfusion protocol activation; blood cell transfusion requirement; surgical control of bleeding requirement and emergent arteriographic embolization. The objective of this study is to demonstrate which of these markers is better to predict hemodynamic evolution of severe trauma patients and might become a guide for resuscitation in the future.

ELIGIBILITY:
Inclusion Criteria:

* Pre-hospital Priority 0 protocol activation:
* Glasgow coma scale < 14
* Systolic blood pressure < 90 mmHg
* Respiratory rate < 10 or > 29 breaths per minute
* Absent peripheral pulses
* Pre-hospital Priority 1 protocol activation:
* All penetratin injuries to head, neck, torso and extremities proximal to elbow and knee
* Flail chest
* Two or more proximal long-bone fractures
* Crushed, degloved or mangled extremity
* Amputation proximal to wrist and ankle
* Pelvic fracture
* Open or depressed skull fracture
* Paralysis

Exclusion Criteria:

* Hospitalization < 24 hours ( transport of the patient to an other trauma center)
* Patients transported from an other hospital (first hours of medical support done elsewhere)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Severe trauma patients admitted at Corporacio Sanitaria Parc Tauli
Sampling Method: Non-Probability Sample
Enrollment: 66 (Actual)
Dates: Start 2016-05; Primary Completion 2019-03-26 (Actual); Study Completion 2019-03-26 (Actual)

PRIMARY OUTCOMES:
Mortality | Through study completion, an average of 1-2 years
  Death of the patient

SECONDARY OUTCOMES:
Multiple organ dysfunction (Multiple Organ Dysfunction Score) | Through study completion, an average of 1-2 years
  Marshall's score (MODS Score) consist on the analysis of 6 systems through different descriptors, those descriptors include: a) the respiratory system (pO2/FIO2 ratio); b) the renal system (serum creatinine concentration); c) the hepatic system (serum bilirrubine concentration); d) the hematologic system (platelet count); and e) the central nervous system (Glasgow Coma Scale); and f) the cardiovascular system (pressure adjusted heart rate). The cardiovascular system descriptor is calculated as the product of the heart rate and the ratio of central venous pressure to mean arterial pressure. All these descriptors will be measured during the first 24h from hospital admission.
Blood cell transfusion | Through study completion, an average of 1-2 years
  Need for blood cell transfusion for patients
Activation of the Massive blood transfusion protocol | At hospital admission
  Need for massive transfusion protocol activation on patients with suspicion of active bleeding
Surgical intervention for bleeding control | Through study completion, an average of 1-2 years
  Need for surgical control on patients with active bleeding
Arteriographic embolization for bleeding control | Through study completion, an average of 1-2 years
  Need for arteriographic embolization on patients with active bleeding

OTHER OUTCOMES:
Hospital stay | Through study completion, an average of 1-2 years
  Number of days that the patient remains in hospital
Intensive care unit stay | Through study completion, an average of 1-2 years
  Number of days that the patient remains in the intensive care unit

CONTACTS AND LOCATIONS:
Overall Officials: Andrea Campos-Serra, MD, Principal Investigator — Corporacion Sanitaria Parc Tauli; Salvador Navarro-Soto, MD, PhD, Study Director — Corporacion Sanitaria Parc Tauli; Sandra Montmany-Vioque, MD, PhD, Study Director — Corporacion Sanitaria Parc Tauli
Locations (1):
- Corporacion Sanitaria Parc Tauli, Sabadell, Barcelona, Spain

REFERENCES:
- [Derived] Campos-Serra A, Mesquida J, Montmany-Vioque S, Rebasa-Cladera P, Barquero-Lopez M, Cidoncha-Secilla A, Llorach-Perucho N, Morales-Codina M, Puyana JC, Navarro-Soto S. Alterations in tissue oxygen saturation measured by near-infrared spectroscopy in trauma patients after initial resuscitation are associated with occult shock. Eur J Trauma Emerg Surg. 2023 Feb;49(1):307-315. doi: 10.1007/s00068-022-02068-w. Epub 2022 Sep 2. PMID 36053289